CLINICAL TRIAL: NCT04693182
Title: Towards a Sustainable Work Force in the Healthcare Sector for the 21st Century: Health-promoting Work Schedules (HeWoS)
Brief Title: Health Promoting Work Schedules: The Effect of Abolishing Quick Returns
Acronym: HeWoS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 303671
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Sick Leave; Insomnia; Shift-Work Sleep Disorder; Psychological Distress; Work Accident; Turnover Intention; Work-family Spillover; Fatigue; Health, Subjective
Keywords: Sick leave, sickness absence, shift work, quick returns
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Circadian Rhythm; Fatigue

STUDY DESIGN:
Intervention Model Description: A parallel-group cluster RCT in a target sample of more than 4000 healthcare workers at Haukeland University Hospital in Norway will be conducted. More than 70 hospital units will be assessed for eligibility and randomized to a work schedule without quick returns for six months or continue with a schedule that maintains quick returns
Who Masked: Outcomes Assessor
Masking Description: All statistical analyses will be done by a researcher who is masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With quick returns (No Intervention): The control condition in this trial implies that employees maintain the same number of quick returns as in previous years for the six-month intervention period. Hospital units in the control group are not expected to experience any increase in the number of quick returns.
- Without quick returns (Experimental): The intervention entails implementing a shift schedule which abolishes quick returns for a six-month intervention period. The number of quick returns in the various hospital units in this trial varies from 329-2356 per year. The intervention means that this number is abolished or reduced as much as possible. For practical reasons it is reasonable to expect that for many of the units it may be a matter of reducing rather than completely abolishing quick returns, as ensuring adequate staffing (e.g., due to sickness absence), often on short-notice make it impossible to comply with the rule of avoiding quick returns. The human resources department at the hospital assisted shift planners in scheduling shift schedules without quick returns.
  Interventions: Other: Shift schedule without quick returns

INTERVENTIONS:
Other: Shift schedule without quick returns — The intervention entails implementing a shift schedule which abolishes or substantially reduces the number of quick returns (less than 11 hours of rest between two shifts) for a six-month intervention period.
  Arms: Without quick returns

SUMMARY:
Introduction In shift work, quick returns refer to transitions between two shifts with less than 11 hours available rest time. Twenty-three per cent of employees in European countries reported having quick returns. Quick returns are related to short sleep duration, fatigue, sleepiness, work-related accidents, and sickness absence. The present study is the first randomized controlled trial (RCT) to investigate the effect of a work schedule without quick returns for six months, compared to a work schedule that maintains quick returns during the same time frame.

Methods and analysis A parallel-group cluster RCT in a target sample of more than 4000 healthcare workers at Haukeland University Hospital in Norway will be conducted. More than 70 hospital units will be assessed for eligibility and randomized to a work schedule without quick returns for six months or continue with a schedule that maintains quick returns. The primary outcome is objective records of sickness absence; secondary outcomes are questionnaire data (n ≈ 4000 invited) on sleep and functioning, physical and psychological health, work-related accidents, and turnover intention. For a subsample, sleep diaries and objective sleep registrations with radar technology (n ≈ 50) will be collected.

Ethics and dissemination The study protocol was approved by the Regional Committee for Medical and Health Research Ethics in Western Norway (2020/200386). Findings from the trial will be disseminated in peer-reviewed journals and presented at national and international conferences. Exploratory analyses of potential mediators and moderators will be reported. User-friendly outputs will be disseminated to relevant stakeholders, unions and other relevant societal groups.

DETAILED DESCRIPTION:
Aims This is a two-arm cluster randomized controlled trial that assesses the consequences of a shift work schedule without quick returns for six months, compared to a schedule that include quick returns. First, we will examine any differential change in sickness absence, during the six-month intervention period. Second, we will examine if there are differential changes in sleep and functioning, physical and mental health, work-related accidents, and turnover intention, among others. Third, we will investigate if individual characteristics associated with shift work tolerance including sex, age, personality and subjectively reported sleep need will moderate the negative effects of quick returns on the primary and secondary outcomes. Finally, the study will investigate if individual factors like satisfaction with work schedule, job satisfaction, job engagement and work-family interference will moderate the negative effects of quick returns on the primary and secondary outcomes.

Research design A cluster randomized controlled trial comparing a work schedule abolishing quick returns (intervention) with that of a work schedule maintaining a normal amount of quick returns (control) will be conducted. The clusters represent hospital units that are randomly selected to receive (or not receive) the intervention. 'Normal amount of quick returns' refer to that which is the common practice at the respective hospital unit in recent years (i.e., when no explicit changes have been made to the work schedule), which means that the total number of quick returns at the unit will vary from 329-2356 per year. The hospital units were randomized to one of the two conditions in September 2020, of which the autumn of 2020 was spent planning the shift schedule for 2021 (i.e., removing quick returns for the intervention group and leaving quick returns untouched for the control group), with the intervention period commencing from February/March 2021 for most units. The intervention period in this study is six calendar months. Most units in this trial start the intervention period in February/March 2021, but some units will, for practical reasons, start the intervention period in the second half of the rotation year, i.e. from August/September 2021 or later.

The primary outcome is sickness absence retrieved from the local records kept by the hospital (including short- and long-term sick leave). The baseline measurements will be sickness absence from the year preceding the intervention, which for each individual participant will be matched on duration and season to that of the intervention period. Sickness absence data will be retrieved from the local records kept by the hospital (Vedaa, Pallesen et al. 2017). This record includes information about the date of any absence of the individual employee, implying that it includes information about both short- and long-term sickness absence. Further, these data include information on whether the absence is self-certified or whether it is certified by a physician, whether the absence is due to a sick child of whom the employee has caretaker responsibility of, and whether the absence is due to COVID-19 related issues (e.g., quarantine). The use of register data will not require individual consent. However, a consent-based part of the trial will also be conducted, in which secondary outcome measures will be collected via questionnaire at baseline and six-month follow-up. All employees (n ≈ 4000) at the randomized units will be asked to complete a digital questionnaire made available via the hospital's internal website. Baseline assessment will occur prior to the intervention period, and follow-up assessment will occur towards the end of the intervention period. A subsample (n ≈ 50) will be asked to objectively record their sleep with advanced radar technomogy (Somnofy™) and subjectively with sleep diaries for ≥1 week at the baseline and follow-up assessments, respectively.

Participants and procedure Recruitment This trial is carried out in close collaboration with the human resources department at Haukeland University Hospital. All hospital care units that have 24-hour staffing at the hospital will be randomized, in which all healthcare workers working shifts will be included, with the exception of physicians. Physicians will not be included since they often have a different shift schedule and compensation scheme compared to the other occupational groups. Hereinafter, 'all employees' refer to all healthcare workers engaged in shift work at the randomised hospital units, with the exception of physicians. All employees (n ≈ 4000) at the randomized hospital units will be asked to complete a questionnaire prior to and at the end of the intervention period. Recruitment for this part of the trial will take place via the hospital's internal website. Researchers and human resources personnel at the hospital will attend staff meetings at all included units to inform about the research project and encourage participation. A subsample of n ≈ 50 randomly selected employees (evenly distributed from the intervention and the control units) will be recruited for the sleep monitoring section of the trial.

Randomisation and masking The randomization in this trial occurred at the cluster level, in which hospital units constituted the clusters. Hospital units can vary in terms of how much staff they need over the 24-hour day, hence, the work schedule and the occurrence of, for example, quick returns and night shifts can vary across the units. Similar units were therefore grouped together based on the fact that they shared some attributes or characteristics. Then a stratified randomization was performed to the two study conditions in a 1: 1 ratio. One subgroup could, for example, consist of units with emergency functions, another with intensive care functions, one with mental health care, and one with maternity care, etc. In total we had 10 strata and the sizes of each stratum varied between 2 and 19 hospital units. The randomization list for each stratum was generated by the online randomization webpage, www.randomization.com, and the list for each stratum was saved.

It is not possible for participants to be blinded to the group to which they are assigned. However, statistical analyses will be done by a researcher who is masked to group allocation.

Sample size In this trial, all available hospital units at Haukeland University Hospital with healthcare workers who work rotating shifts will be assessed for eligibility. This includes 76 units and 4260 healthcare workers. Based on previous published data5 we have calculated that a total of 2028 participants is sufficient to reveal a difference in days of sick leave of 0.9 and 1.25 with an ICC of 0.1 and an average size of the units of 52 (calculation made in: StataCorp. 2015).33 Thus, with the planned recruitment strategy (i.e., invite >70 units and >4000 healthcare workers) we expect to exceed this number and be well within the number of participants required for the primary outcome variable.

Data analysis plan All analyses will be conducted based on the intention-to-treat population, unless otherwise stated. To examine the effects of a shift schedule abated of quick returns on primary and secondary outcomes, the observed rates or scores will be analysed by means of latent growth models (or other equivalent models such as generalized linear mixed models). The observed rates or scores before and during the intervention period will be modelled by a random intercept and a fixed slope. The effect of the intervention will be estimated by using the group variable (intervention vs. control) as a predictor of the slope. Between-group effect sizes (Cohen's d) will be calculated by dividing the mean difference in estimated change in scores from baseline to the follow-up assessment by the pooled SD at baseline. Robust maximum likelihood will be used as the estimator, providing unbiased estimates under the assumption of data being missing at random,(Enders 2010) which might be partly met through the inclusion of baseline scores to the model. The primary outcome measure in this trial is sickness absence data retrieved from the register at the hospital, in which we expect no missing data. However, it is reasonable to expect some missing data on the secondary outcome measures, as data are collected through questionnaire or via the sleep radar.

As some data for the follow-up questionnaire and sleep radar assessment will be missing not at random, the robustness of the results under the missing-at-random assumption will be tested by sensitivity analyses in which the missing scores at follow-up will be replaced by baseline values for each respective individual. These sensitivity analyses will only be performed on selected variables depending on the focus in the respective article.

The intention-to-treat analyses may be accompanied by selected per-protocol analyses in which we, based on payroll data, define a group that has completely abolished or had a satisfactory reduction in the number of quick returns over the intervention period.

The primary outcome of sick leave will mainly be analysed in terms of the total number of sickness absence days and periods (spells) for a given period before compared to during the intervention period (Vedaa, Pallesen et al. 2017). The models of sickness absence will take into account the zero inflation in this type of data. Other operationalisations of sickness absence might also be considered in accordance with recommendations in the literature (Hensing, Alexanderson et al. 1998). For a further investigation of the sickness absence data, we will consider the use of other models where we treat time differently. For example, we will consider models where we look at the time to the first sick leave episode for the two intervention groups, with a time-dependent covariate for the number of quick returns (ie, a variable that increases by 1 each time the person has a quick return). Another possibility is to say that participants start at "0" every time the person has a quick return, and to measure time from the last quick return to the first subsequent sick leave episode, while adjusting for repeated observations with e.g. robust variance estimate (the non-quick return group will then only be followed from the start of the intervention, given that they in fact have no quick returns). Another option is to set up a model for time from sick leave to return to work.

Since the introduction of a work schedule without quick returns may entail an alternative schedule with an increase in other undesirable characteristics (e.g., more consecutive evening shifts), we will consider conducting analyses that adjust for such characteristics.

Mediator and moderator analyses will be performed for exploratory purposes, based on the basic principle for such analyses in randomised controlled trials as described by others ((e.g., Kraemer, Wilson et al. 2002)). For example, some of the data collected on demographics, sleep-related personality traits (rCTI and MEQ), mental health, among others, can be used to examine factors that may moderate the impact of the intervention.

References

Enders, C. K. (2010). Applied missing data analysis. New York, NY, US, Guilford Press.

Hensing, G., et al. (1998). "How to measure sickness absence? Literature review and suggestion of five basic measures." Scandinavian journal of public health 26: 133-144.

Kraemer, H. C., et al. (2002). "Mediators and moderators of treatment effects in randomized clinical trials." Archives of General Psychiatry 59: 877-883.

Vedaa, Ø., et al. (2017). "Short rest between shift intervals increases the risk of sick leave: a prospective registry study." Occupational and Environmental Medicine 74: 496-501.

ELIGIBILITY:
Inclusion Criteria:

* The unit-level inclusion criteria are that the units should have: 1) healthcare workers (other than physicians) who work rotating shifts, 2) employees who regularly have quick returns in their work schedule, and 3) a new shift rotation year commencing from February/March 2021 (which is the case for most units at Haukeland University Hospital).
* Employees must be healthcare workers at the above-mentioned hospital units.
* Employees must have >50% position.

Exclusion Criteria:

* Exclusion criteria at the unit-level are 1) units have recently (or will in the near future) went through other major organizational changes that may confound the results (this includes during the period from one year before the intervention starts until the intervention period is over) of the trial, or 2) unit's manager or a substantial number of employees strongly oppose participation in the trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Sickness absence | For example, sickness absence in the last three months of the intervention period will be compared with three months the year before the intervention started, matched in terms of season.
  Sickness absence data will be retrieved from the local register at the hospital. Sickness absence will mainly be analysed in terms of the total number of sickness absence days and periods (spells) for a given period before compared to during the intervention period.

SECONDARY OUTCOMES:
Insomnia | Questionnaires are answered before and towards the end of the six-month intervention period
  The Bergen Insomnia Scale
Shift work disorder | Questionnaires are answered before and towards the end of the six-month intervention period
  Shift work disorder will be measured with three standardised questions
Fatigue | Questionnaires are answered before and towards the end of the six-month intervention period
  The Swedish Occupational Fatigue Inventory
Job satisfaction | Questionnaires are answered before and towards the end of the six-month intervention period
  Job satisfaction will be assessed with five items (e.g., "I find real enjoyment in my work") from the Job Satisfaction Index
Mental Health | Questionnaires are answered before and towards the end of the six-month intervention period
  Hopkins symptom checklist - 5
Work-family spillover | Questionnaires are answered before and towards the end of the six-month intervention period
  The Work family Interface Scale developed by Kinnunen, Feldt, Geurts et al. will be used to evaluate the four types of work-family spillover
Work-related negative incidents | Questionnaires are answered before and towards the end of the six-month intervention period
  Work-related negative incidents will be assessed using eight items measuring the number of self-reported work-related accidents, near accidents and dozing off at work or while driving to or from work.
Turnover Intention | Questionnaires are answered before and towards the end of the six-month intervention period
  The Turnover Intention Scale will be measured with the three-item Turnover Intention Scale adapted from Michigan Organizational Assessment Questionnaire
Sleep (subjective and objective) | Sleep is measured with a sleep diary and sleep radar for >7 days before and towards the end of the six-month intervention period.
  Will be measured subjectively with a sleep diary and objectively with a Xethru sensor, a low-powered ultra-wideband radar.
Subjective health complaints | Questionnaires are answered before and towards the end of the six-month intervention period
  Subjective health complaints inventory (only parts of the scale will be used)

OTHER OUTCOMES:
Unwanted / negative effects | Possible negative outcomes of the intervention will be measured after the intervention period.
  We will measure if changed work schedule has led to disturbed sleep, more stress, worry, depression, overall less time for recovery between work periods, problems in work-family balance, disrupted social relationships, poorer psychosocial climate at work, experience of reduced quality of care offered to patients, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Anette Harris, PhD, Principal Investigator — University of Bergen, Norway
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified data that underlie the results reported from the trial described in this protocol will be available to researchers from accredited research institutions. Access to data will be limited to investigators who provide a methodologically sound proposal and will be limited to a specified time period (commencing about 3 months after publication of a respective Article and ending after 5 years). To ensure compliance with the General Data Protection Regulation, data processing must be covered by the European Commission's standard contractual clauses for the transfer of data, which must be signed by the data requesters. Proposals and requests for data access should be directed to the corresponding author of the respective Article. User-friendly output from the trial will be disseminated to stakeholder and other relevant organisations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data that underlie the results reported from the trial described in this protocol will be available to researchers from accredited research institutions. Access to data will be limited to investigators who provide a methodologically sound proposal and will be limited to a specified time period (commencing about 3 months after publication of a respective Article and ending after 5 years).
Access Criteria: To ensure compliance with the General Data Protection Regulation, data processing must be covered by the European Commission's standard contractual clauses for the transfer of data, which must be signed by the data requesters. Proposals and requests for data access should be directed to the corresponding author of the respective Article.

REFERENCES:
- [Derived] Djupedal ILR, Harris A, Svensen E, Lie SA, Wang ALH, Pallesen S, Waage S, Nielsen MB, Sunde E, Bjorvatn B, Holmelid O, Vedaa O. Shift Schedule With Fewer Short Daily Rest Periods and Sickness Absence Among Health Care Workers: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2531568. doi: 10.1001/jamanetworkopen.2025.31568. PMID 40952742
- [Derived] Djupedal ILR, Harris A, Svensen E, Pallesen S, Waage S, Nielsen MB, Sunde E, Bjorvatn B, Holmelid O, Vedaa O. Effects of a work schedule with abated quick returns on insomnia, sleepiness, and work-related fatigue: results from a large-scale cluster randomized controlled trial. Sleep. 2024 Jul 11;47(7):zsae086. doi: 10.1093/sleep/zsae086. PMID 38581363
- [Derived] Vedaa O, Djupedal ILR, Svensen E, Waage S, Bjorvatn B, Pallesen S, Lie SA, Nielsen M, Harris A. Health-promoting work schedules: protocol for a large-scale cluster randomised controlled trial on the effects of a work schedule without quick returns on sickness absence among healthcare workers. BMJ Open. 2022 Apr 15;12(4):e058309. doi: 10.1136/bmjopen-2021-058309. PMID 35428642
- See also: Link to information letter to participants — https://www.uib.no/fg/sc/141586/informasjon-til-deltagere
- See also: Link to the study website — https://www.uib.no/fg/sc/141585/effekt-av-en-arbeidsplan-uten-kort-hviletid